CLINICAL TRIAL: NCT04661826
Title: ONCOFID-P-B (PACLITAXEL-HYALURONIC ACID) in the Intravescical Therapy of Patients With Non-muscle Invasive Cancer of the Bladder. A Phase II Marker Lesion. STUDY
Brief Title: ONCOFID-P-B in the Intravescical Therapy of Patients With Non-muscle Invasive Cancer of the Bladder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R39-09-01
Record Dates: First submitted 2020-12-02; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Non-Invasive Papillary Carcinoma of Bladder
Keywords: paclitaxel; bladder cancer; hyaluronic acid
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncofid-P-B (Experimental): Oncofid-P-B will be administered once a week for 6 weeks in the first treatment phase and once a month for 6 months followed by other 6 months in the second maintenance phase
  Interventions: Drug: Oncofid-P-B

INTERVENTIONS:
Drug: Oncofid-P-B — Paclitaxel - Hyaluronic Acid 600 mg - Solution for intravesical administration.

SUMMARY:
The purpose of the study is to assess, at control visit (V8), the ablative activity of intravesical administration of Oncofid-P-B on a papillary marker tumor on patients suffering from multiple primary and recurrent Ta G1-G2 papillary cancer of the bladder after 6 weeks of weekly study drug administration, through number and percentage of patients with Complete Response.

DETAILED DESCRIPTION:
This study will investigate the preliminary activity of Oncofid-P-B administered by intravescical route at the Recommended Dose of 600 mg, once a week, for six weeks evaluating the ablative activity on a papillary marker tumor in patients suffering from non-muscle invasive cancer of the bladder. When a patient will present a Complete Response at the end of the six weekly administration of Oncofid-P-B , he/she can enter a second phase of the study defined maintenance phase. During this phase, the patients will be treated with the study drug administered by intravesical infusion once a month for 2 cycles of treatment with the duration of 6 months separated by a period during which study drug will not be administered, due to the necessity to perform histological evaluation of efficacy. This scheme will follow a clinical usual approach for the maintenance treatment of patients suffering from non-muscle invasive cancer of the bladder.

Complete Response is defined as follows: complete disappearance of the marker lesion, as confirmed by negative post-treatment cystoscopy including a biopsy at the marker lesion site and the absence of new tumors at other site and negative cytology.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged > 18 years, women in menopause (defined as surgically sterile or one year postmenopausal);
* Cytological or histological diagnosis of bladder cancer;
* Multiple primary or recurrent Ta G1-G2 papillary cancer;
* ECOG Performance Status 0 to 1;
* Adequate bone marrow function: neutrophils ≥1.5 103/mL; platelet count ≥100 103/ mm3; Hb ≥ 10 g/dL;
* Written informed consent;
* Willing and able to comply with the protocol for the duration of the study.

Exclusion Criteria:

* Hypersensitivity to Paclitaxel or one of its constituents;
* T1 papillary cancer or muscle-invasive disease (T2-T4) ;
* Previous or concomitant tumor of the upper urinary tract, of the prostatic urethra, CIS;
* Any other malignancy diagnosed within 3 years of study entry (except basal or squamous cell skin cancers or non-invasive cancer of the cervix);
* Presence of significant urologic disease interfering with intravesical therapy;
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening or concurrent treatment with other experimental drugs;
* Other chemotherapy or radiotherapy within four weeks of study entry;
* Previous intravesical immunotherapy or chemotherapy less than 3 months before study entry;
* Bladder capacity less than 300 mL;
* Renal and hepatic function values exceeding 2 times the upper normal value;
* Severe cardiovascular diseases considered a contraindication to intravesical treatment;
* Pregnant, lactating or childbearing potential aged women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2015-07-29 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
CR at control visit (V8) after intravescical administration of Oncofid-P-B on a papillary marker tumor. | Visit 8 will be performed 2-4 weeks after the last treatment visit (Visit 7)
  Rate of complete response, estimated at V8, after 6 weeks of weekly study drug administration: number and percentage of patients with complete response. Complete response is defined as follows: complete disappearance of the marker lesion, as confirmed by negative post-treatment cystoscopy including a biopsy at the marker lesion site and the absence of new tumors at other sites and negative cytology.

SECONDARY OUTCOMES:
Time to relapse after Oncofid-P-B instillation during the maintenance phase. | The second treatment maintenance phase constituted by 2 treatment periods with a duration of 6 months each (comprehensively considered equal to 52 weeks).
  Time to relapse after Oncofid-P-B instillation during the maintenance phase.
Number of patients with relapse within V 22. | The second treatment maintenance phase constituted by 2 treatment periods with a duration of 6 months each (comprehensively considered equal to 52 weeks).
  Number of patients with relapse within V 22.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0" | The second treatment maintenance phase constituted by 2 treatment periods with a duration of 6 months each (comprehensively considered equal to 52 weeks).
  Treatment-Related Adverse Events as Assessed by CTCAE v4.0" with Oncofid-P-B given by intravesical instillation.

CONTACTS AND LOCATIONS:
Locations (14):
- Germany (3):
  - Klinik und Poliklinik für Urologie, Kinderurologie und Onkologische Urologi, Essen
  - Urologische Klinik und Poliklinik - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Praxisklinik Urologie Rhein-Ruhr, Mülheim
- Italy (5):
  - A.O.Universitaria - Ospedale Consorziale Policlinico di Bari - Urologia - Dipartimento d'Emergenza e dei Trapianti di Organi, Bari
  - A.O. Spedali Civili di Brescia - Dipartimento di Urologia, Brescia
  - Azienda Ospedaliera Universitaria di Pisa - U.O. Urologia Universitaria, Pisa
  - Policlinico A.Gemelli - Università Cattolica del Sacro Cuore - Dipartimento di Scienze Chirurgiche - Clinica Urologica, Roma
  - A.O.Città della Salute e della Scienza di Torino - Ospedale Molinette Dipartimento di Urologia I, Torino
- Spain (6):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital del Henares, Coslada, Madrid
  - Tenerife Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Instituto Valenciano de Oncologià, Valencia